CLINICAL TRIAL: NCT00588926
Title: Changes of the Neuronal Activity in the Subthalamic Nucleus Under Remifentanil Sedation During Stereotactic Electrode Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Dan Eimerl, M.D., Dept. Anesthesiology, Hadassah Medical Center, Jerusalem, Israel.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 221107-hmo-ctil
Record Dates: First submitted 2007-12-30; First posted 2008-01-09 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Movement Disorders; Effect of Remifentanil
Keywords: Deep Brain Stimulation; Movement Disorders; Remifentanil; Sedation; Basal Ganglia electrical activity
MeSH Terms: conditions — Movement Disorders | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): The patients get a period of sedation with remifentanil, before, during and after which, the changes in the electrical activity of the Basal Ganglia is recorded.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — After the mapping electrode is in situ, recording of baseline electrical activity is done for two-three minutes and an infusion of Remifentanil, 0.1 microgram per kilogram per minute is started. This procedure continues for a few minutes until the patient is sedated and then the infusion is stopped and the patient allowed to recover. The recordings continue during the whole procedure.

SUMMARY:
Deep brain stimulation is commonly used for the treatment of movement disorders. Electrode positioning is usually performed under local anesthesia in fully awake patients. The procedure is uncomfortable to the patients who has to remain motionless during the whole surgery. Previous reports of electrode positioning under general anesthesia was found to be less accurate. This result was probably due to the effect of the anesthetics on the electrical activity of the basal ganglia.

The purpose of this study is to detect possible changes in the electrical activity of the basal ganglia related to remifentanil sedation. electrical activity of single neurons will be recorded before, during and after sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with movement disorder, who are candidates for implantation of deep brain stimulation electrode.

Exclusion Criteria:

* Suspected difficult intubation
* history of sleep apnea
* known allergy for remifentanil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)

PRIMARY OUTCOMES:
Electrical activity in the basal ganglia | During the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Dan Eimerl, MD, Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Derived] Benady A, Zadik S, Eimerl D, Heymann S, Bergman H, Israel Z, Raz A. Sedative drugs modulate the neuronal activity in the subthalamic nucleus of parkinsonian patients. Sci Rep. 2020 Sep 3;10(1):14536. doi: 10.1038/s41598-020-71358-3. PMID 32884017